CLINICAL TRIAL: NCT01764386
Title: A Multicenter, Randomized, Open-Label, Controlled, Method-of-Use Study Assessing the Effect of Naltrexone Sustained Release (SR)/Bupropion SR on Body Weight and Cardiovascular Risk Factors in Overweight and Obese Subjects (The Ignite Study)
Brief Title: Method-of-Use Study Assessing the Effect of Naltrexone Sustained Release (SR)/ Bupropion SR on Body Weight and Cardiovascular Risk Factors in Overweight and Obese Subjects
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Orexigen Therapeutics, Inc (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NB-404
Record Dates: First submitted 2013-01-04; First posted 2013-01-09 (Estimated); Results first posted 2015-11-26 (Estimated); Last update posted 2015-12-29 (Estimated); Status verified 2015-11

CONDITIONS: Obesity; Overweight
Keywords: obesity, overweight
MeSH Terms: conditions — Obesity; Overweight

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- NB + CLI (Experimental): Naltrexone SR 32 mg/Bupropion SR 360 mg/day (NB) with comprehensive lifestyle intervention (CLI)
  Interventions: Drug: NB; Behavioral: CLI
- Usual Care (Other): Usual Care (self-directed lifestyle intervention)
  Usual Care: Usual Care was a self-directed lifestyle intervention in which subjects were given calorie targets, instructions to increase exercise, and a pamphlet about weight loss by study site staff.
  Interventions: Behavioral: Usual Care

INTERVENTIONS:
Drug: NB — Naltrexone SR 32 mg/Bupropion SR 360 mg (NB) in combination tablets (daily dosage)
  Arms: NB + CLI
Behavioral: CLI — The Comprehensive Lifestyle Intervention (CLI) program includes telephone counseling, internet education, goal setting, and online tracking tools.
  Arms: NB + CLI
Behavioral: Usual Care — Usual Care is a self-directed lifestyle intervention program
  Arms: Usual Care

SUMMARY:
The purpose of this Phase 3b study is to assess the effects of combination therapy with naltrexone SR/bupropion SR (NB) used in conjunction with a comprehensive lifestyle intervention (CLI) and in a manner consistent with its intended use after marketing approval, on body weight and cardiovascular risk factors compared to the effects of Usual Care in subjects who are overweight with dyslipidemia and/or controlled hypertension or obese. Subjects in the NB and CLI group are required to undergo an evaluation to continue treatment at Week 16. Subjects are to be discontinued from full participation if they do not lose at least 5% of their body weight relative to baseline and/or are experiencing sustained increases in blood pressure (systolic or diastolic) of ≥10 mmHg above baseline. At Week 26, subjects originally assigned to Usual Care switch to treatment with NB and CLI, and subjects assigned to NB and CLI continue treatment for the duration of the study (78-weeks treatment period).

ELIGIBILITY:
Inclusion Criteria:

* Female or male, 18 to 60 years old
* Body mass index (BMI) ≥30 kg/m2 and ≤45 kg/m2 for subjects with uncomplicated obesity, or BMI ≥27 kg/m2 and ≤45 kg/m2 for subjects with dyslipidemia and/or controlled hypertension

Exclusion Criteria:

* History of type 1 or type 2 diabetes mellitus diagnosis
* Myocardial infarction within 6 months prior to screening
* Angina pectoris Grade III or IV as per the Canadian Cardiovascular Society grading scheme
* Clinical history of large vessel cortical strokes, including ischemic and hemorrhagic strokes (i.e., transient ischemic attack is not exclusionary)
* History (within the last 20 years) of seizures, cranial trauma, bulimia, anorexia nervosa, or other conditions that predispose subjects to seizures
* Past or planned surgical or device intervention (e.g., gastric banding) for obesity
* Chronic use or positive screen for opioids
* Regular use of tobacco products

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 242 (Actual)
Dates: Start 2013-02; Primary Completion 2014-09 (Actual); Study Completion 2014-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Senior Vice President, Head of Global Development, Study Director — Orexigen Therapeutics, Inc
Locations (15):
- United States (15):
  - Radiant Research, Denver, Colorado
  - Radiant Research, Inc., St Louis, Missouri
  - PMG Research of Raleigh, Cary, North Carolina
  - PMG Research of Winston-Salem, Hickory, North Carolina
  - PMG Research of Raleigh, Raleigh, North Carolina
  - PMG Research of Salisbury, Salisbury, North Carolina
  - PMG Research of Wilmington, LLC, Wilmington, North Carolina
  - Radiant Research-Akron, Akron, Ohio
  - Radiant Research, Inc., Columbus, Ohio
  - Radiant Research, Anderson, South Carolina
  - Radiant Research, Greer, Greer, South Carolina
  - PMG Research of Charleston, Mt. Pleasant, South Carolina
  - PMG Research of Bristol, Bristol, Tennessee
  - Radiant Research Dallas-North, Dallas, Texas
  - Radiant Research, SLC, Salt Lake City, Utah

REFERENCES:
- [Derived] Halseth A, Shan K, Walsh B, Gilder K, Fujioka K. Method-of-use study of naltrexone sustained release (SR)/bupropion SR on body weight in individuals with obesity. Obesity (Silver Spring). 2017 Feb;25(2):338-345. doi: 10.1002/oby.21726. Epub 2016 Dec 27. PMID 28026920

RESULTS

PARTICIPANT FLOW:
Groups:
- NB + CLI: Naltrexone SR 32 mg/Bupropion SR 360 mg/day (NB) with Comprehensive Lifestyle Intervention (CLI)
  NB: Naltrexone SR 32 mg/Bupropion SR 360 mg (NB) in combination tablets (daily dosage)
  CLI: The Comprehensive Lifestyle Intervention (CLI) program included telephone counseling, internet education, goal setting, and online tracking tools.
  The Controlled Treatment Period was from Day 1 to Week 26. The Uncontrolled Treatment Period was from Week 26 to Week 78. At the end of the Controlled Treatment Period (Week 26), subjects assigned to NB+CLI continued with NB+CLI for the duration of the study (Week 78).
- Usual Care: Usual Care (self-directed lifestyle intervention)
  Usual Care: Usual Care was a self-directed lifestyle intervention in which subjects were given calorie targets, instructions to increase exercise, and a pamphlet about weight loss by study site staff.
  The Controlled Treatment Period was from Day 1 to Week 26. The Uncontrolled Treatment Period was from Week 26 to Week 78. At the end of the Controlled Treatment Period (Week 26), subjects assigned to Usual Care were switched to NB+CLI for the duration of the study (Week 78).
Period: Controlled Treatment Period (CTP)
Arm/Group | NB + CLI | Usual Care
Started | 153 | 89
Completed | 71 (Completed the 26-week Controlled Treatment Period.) | 82 (Completed the 26-week Controlled Treatment Period.)
Not Completed | 82 | 7
Not completed — Adverse Event | 35 | 0
Not completed — Wk 16 Efficacy and BP Criteria | 32 | 0
Not completed — Lost to Follow-up | 9 | 5
Not completed — Withdrawal of Consent,Protocol Deviation | 6 | 2
Period: Uncontrolled Treatment Period (UTP)
Arm/Group | NB + CLI | Usual Care
Started | 71 | 81 (One subject completed the 26-week CTP, but did not continue in the UTP.)
Completed 52 Weeks | 61 | 35
Completed | 55 (Completed the 78-week study.) | 28 (Completed the 78-week study.)
Not Completed | 16 | 53
Not completed — Adverse Event | 2 | 13
Not completed — Wk 42 Efficacy and BP Criteria | 0 | 26
Not completed — Lost to Follow-up | 9 | 9
Not completed — Withdrawal of Consent,Protocol Deviation | 5 | 5

BASELINE CHARACTERISTICS:
Population: Baseline analysis was based on the Intent-to-Treat (ITT) population which comprised all subjects randomized to NB + CLI who received at least 1 dose of study medication and all subjects randomly assigned to Usual Care who received their baseline lifestyle intervention program instruction.
Groups:
- NB + CLI: Naltrexone SR 32 mg/Bupropion SR 360 mg/day (NB) with Comprehensive Lifestyle Intervention (CLI)
  NB: Naltrexone SR 32 mg/Bupropion SR 360 mg (NB) in combination tablets (daily dosage)
  CLI: The Comprehensive Lifestyle Intervention (CLI) program included telephone counseling, internet education, goal setting, and online tracking tools.
- Total: Total of all reporting groups
Arm/Group | NB + CLI | Usual Care | Total
Number analyzed (Participants) | 153 | 89 | 242
Age, Continuous [Mean (Standard Deviation); unit: years] | 46.1 (9.66) | 47.0 (9.98) | 46.5 (9.77)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 125 | 77 | 202
  Male | 28 | 12 | 40
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 4 | 5 | 9
  Not Hispanic or Latino | 149 | 84 | 233
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 1 | 1
  Asian | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 28 | 24 | 52
  White | 124 | 64 | 188
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 153 | 89 | 242
Weight [Mean (Standard Deviation); unit: kg] | 101.4 (15.09) | 100.2 (16.58) | 100.9 (15.63)
Baseline BMI [Mean (Standard Deviation); unit: kg/m^2] | 36.33 (4.200) | 36.26 (4.369) | 36.31 (4.254)

OUTCOME MEASURES:

1. Primary Outcome: Percent Change in Body Weight From Baseline (Day 1) to Week 26
Time Frame: Baseline to Week 26
Population: The Week 26 Per Protocol (PP) population comprised subjects from the mITT population (i.e., ITT subjects with their Week 2 study visit, with baseline [BL] and at least 1 post-BL body weight measured) who had completed the study through Week 26 in compliance with the protocol. Subjects in the NB + CLI group had to be on study medication at Week 26.
Measure: Least Squares Mean (Standard Error); unit: percent change in body weight
Arm/Group | NB + CLI | Usual Care
Number analyzed (Participants) | 71 | 82
percent change in body weight | -9.46 (0.54) | -0.94 (0.49)
Statistical Analysis 1: Comparison: NB + CLI vs Usual Care; Test type: Superiority or Other; p < 0.0001, ANCOVA; Mean Difference (Net) = -8.52, 95% CI 2-sided [-9.88 to -7.15]

2. Secondary Outcome: Percentage of Subjects Achieving a Loss of at Least 5% of Baseline Body Weight at Week 26
Time Frame: Baseline to Week 26
Population: as for outcome 1
Measure: Number; unit: percentage of participants
Arm/Group | NB + CLI | Usual Care
Number analyzed (Participants) | 71 | 82
percentage of participants | 84.5 | 12.2
Statistical Analysis 1: Comparison: NB + CLI vs Usual Care; Test type: Superiority or Other; p < 0.0001, Regression, Logistic; Odds Ratio (OR) = 44.0, 95% CI 2-sided [16.6 to 116.3]

3. Secondary Outcome: Percentage of Subjects Achieving a Loss of at Least 10% of Baseline Body Weight at Week 26
Time Frame: Baseline to Week 26
Population: as for outcome 1
Measure: Number; unit: percentage of participants
Arm/Group | NB + CLI | Usual Care
Number analyzed (Participants) | 71 | 82
percentage of participants | 42.3 | 3.7
Statistical Analysis 1: Comparison: NB + CLI vs Usual Care; Test type: Superiority or Other; p < 0.0001, Regression, Logistic; Odds Ratio (OR) = 21.4, 95% CI 2-sided [6.0 to 76.7]

4. Secondary Outcome: Percentage of Subjects Achieving a Loss of at Least 15% of Baseline Body Weight at Week 26
Time Frame: Baseline to Week 26
Population: as for outcome 1
Measure: Number; unit: percentage of participants
Arm/Group | NB + CLI | Usual Care
Number analyzed (Participants) | 71 | 82
percentage of participants | 12.7 | 0.0

5. Secondary Outcome: Absolute Change in Body Weight From Baseline to Week 26
Time Frame: Baseline to Week 26
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: kg
Arm/Group | NB + CLI | Usual Care
Number analyzed (Participants) | 71 | 82
kg | -9.7 (0.56) | -1.0 (0.51)
Statistical Analysis 1: Comparison: NB + CLI vs Usual Care; Test type: Superiority or Other; p < 0.0001, ANCOVA; Mean Difference (Net) = -8.65, 95% CI 2-sided [-10.07 to -7.24]

6. Secondary Outcome: Change in Waist Circumference From Baseline to Week 26
Time Frame: Baseline to Week 26
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: cm
Arm/Group | NB + CLI | Usual Care
Number analyzed (Participants) | 71 | 82
cm | -6.96 (0.705) | -1.64 (0.659)
Statistical Analysis 1: Comparison: NB + CLI vs Usual Care; Test type: Superiority or Other; p < 0.0001, ANCOVA; Mean Difference (Net) = -5.32, 95% CI 2-sided [-7.14 to -3.50]

7. Secondary Outcome: Change in Fasting Triglycerides From Baseline to Week 26
Time Frame: Baseline to Week 26
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: mg/dL
Arm/Group | NB + CLI | Usual Care
Number analyzed (Participants) | 71 | 82
mg/dL | -13.6 (4.96) | 2.8 (4.63)
Statistical Analysis 1: Comparison: NB + CLI vs Usual Care; Test type: Superiority or Other; p = 0.0019, ANCOVA; Mean Difference (Net) = -16.4, 95% CI 2-sided [-29.5 to -3.3]

8. Secondary Outcome: Change in Fasting Low-density Lipoprotein Cholesterol From Baseline to Week 26
Time Frame: Baseline to Week 26
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: mg/dL
Arm/Group | NB + CLI | Usual Care
Number analyzed (Participants) | 71 | 82
mg/dL | -2.0 (2.20) | -1.9 (2.11)
Statistical Analysis 1: Comparison: NB + CLI vs Usual Care; Test type: Superiority or Other; p = 0.9686, ANCOVA; Mean Difference (Net) = -0.1, 95% CI 2-sided [-5.96 to 5.73]

9. Secondary Outcome: Change in Fasting High-density Lipoprotein Cholesterol From Baseline to Week 26
Time Frame: Baseline to Week 26
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: mg/dL
Arm/Group | NB + CLI | Usual Care
Number analyzed (Participants) | 71 | 82
mg/dL | 4.1 (0.77) | 0.1 (0.73)
Statistical Analysis 1: Comparison: NB + CLI vs Usual Care; Test type: Superiority or Other; p = 0.0001, ANCOVA; Mean Difference (Net) = 4.0, 95% CI 2-sided [1.99 to 6.06]

10. Secondary Outcome: Change in Systolic Blood Pressure From Baseline to Week 26
Time Frame: Baseline to Week 26
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: mm Hg
Arm/Group | NB + CLI | Usual Care
Number analyzed (Participants) | 71 | 82
mm Hg | -4.8 (1.10) | -2.8 (1.02)
Statistical Analysis 1: Comparison: NB + CLI vs Usual Care; Test type: Superiority or Other; p = 0.1706, ANCOVA; Mean Difference (Net) = -2.0, 95% CI 2-sided [-4.9 to 0.9]

11. Secondary Outcome: Change in Diastolic Blood Pressure From Baseline to Week 26
Time Frame: Baseline to Week 26
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: mm Hg
Arm/Group | NB + CLI | Usual Care
Number analyzed (Participants) | 71 | 82
mm Hg | -1.7 (0.83) | -1.3 (0.77)
Statistical Analysis 1: Comparison: NB + CLI vs Usual Care; Test type: Superiority or Other; p = 0.7160, ANCOVA; Mean Difference (Net) = -0.4, 95% CI 2-sided [-2.6 to 1.8]

12. Secondary Outcome: Change in Heart Rate From Baseline to Week 26
Time Frame: Baseline to Week 26
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: bpm
Arm/Group | NB + CLI | Usual Care
Number analyzed (Participants) | 71 | 82
bpm | 1.7 (0.88) | -0.3 (0.82)
Statistical Analysis 1: Comparison: NB + CLI vs Usual Care; Test type: Superiority or Other; p = 0.0913, ANCOVA; Mean Difference (Net) = 2.0, 95% CI 2-sided [-0.3 to 4.3]

13. Secondary Outcome: Change in Fasting Plasma Glucose From Baseline to Week 26
Time Frame: Baseline to Week 26
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: mg/dL
Arm/Group | NB + CLI | Usual Care
Number analyzed (Participants) | 71 | 82
mg/dL | -2.9 (1.04) | 1.6 (0.96)
Statistical Analysis 1: Comparison: NB + CLI vs Usual Care; Test type: Superiority or Other; p = 0.0016, ANCOVA; Mean Difference (Net) = -4.5, 95% CI 2-sided [-7.2 to -1.7]

14. Secondary Outcome: Change Fasting Insulin From Baseline to Week 26
Time Frame: Baseline to Week 26
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: uIU/mL
Arm/Group | NB + CLI | Usual Care
Number analyzed (Participants) | 71 | 82
uIU/mL | -7.5 (0.79) | -3.4 (0.76)
Statistical Analysis 1: Comparison: NB + CLI vs Usual Care; Test type: Superiority or Other; p = 0.0004, ANCOVA; Mean Difference (Net) = -4.1, 95% CI 2-sided [-6.2 to -2.0]

15. Secondary Outcome: Change in Homeostasis Model Assessment-insulin Resistance (HOMA-IR) From Baseline to Week 26
Description: HOMA-IR is an insulin sensitivity index that is calculated as HOMA-IR = (Glucose * Insulin) / 405, where glucose is in mass units (mg/dL) and insulin is in µIU/mL. Higher values indicate lower insulin sensitivity.
Time Frame: Baseline to Week 26
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | NB + CLI | Usual Care
Number analyzed (Participants) | 71 | 82
units on a scale | -2.0 (0.20) | -0.8 (0.19)
Statistical Analysis 1: Comparison: NB + CLI vs Usual Care; Test type: Superiority or Other; p = 0.0003, ANCOVA; Mean Difference (Net) = -1.2, 95% CI 2-sided [-1.7 to -0.7]

16. Secondary Outcome: Change in Patient-reported Binge Eating Scale (BES) Total Scores From Baseline to Week 26
Description: The BES is a 16-item questionnaire that identifies different levels of binge-eating severity, with total scores ranging between 0-46. BES scores were categorized as follows: None = Scores ≤17 indicated no significant binge eating, Moderate = scores from 18 to 26 (inclusive), Severe = scores ≥27 indicated severe levels of binge eating.
Time Frame: Baseline to Week 26
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | NB + CLI | Usual Care
Number analyzed (Participants) | 71 | 82
units on a scale | -6.8 (0.72) | 1.1 (0.67)
Statistical Analysis 1: Comparison: NB + CLI vs Usual Care; Test type: Superiority or Other; p < 0.0001, ANCOVA; Mean Difference (Net) = -7.9, 95% CI 2-sided [-9.8 to -6.0]

17. Secondary Outcome: Change in Patient-reported Arizona Sexual Experiences Scale (ASEX) Total Scores From Baseline to Week 26
Description: Arizona Sexual Experiences (ASEX) scale is a 5-item rating scale that quantifies sex drive, arousal, vaginal lubrication/penile erection, ability to reach orgasm, and satisfaction from orgasm. Possible total scores range from 5 to 30, with the higher scores indicating more sexual dysfunction.
Time Frame: Baseline to Week 26
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | NB + CLI | Usual Care
Number analyzed (Participants) | 71 | 82
units on a scale | -2.2 (0.36) | -0.1 (0.34)
Statistical Analysis 1: Comparison: NB + CLI vs Usual Care; Test type: Superiority or Other; p < 0.0001, ANCOVA; Mean Difference (Net) = -2.1, 95% CI 2-sided [-3.1 to -1.1]

18. Secondary Outcome: Change in Patient-reported Impact of Weight on Quality of Life-Lite Questionnaire (IWQOL-Lite) Total Score From Baseline to Week 26
Description: Impact of Weight on Quality of Life-Lite Questionnaire (IWQOL-Lite) is a self-reported assessment of perceived effect of weight on quality of life. It consists of 31 items organized in 5 domains (physical function, self-esteem, sexual life, public distress and work). IWQOL-Lite total score is based on a scale from 0 to 100, with 0 representing the poorest and 100 the best quality of life and where a score of 71-79 indicates moderate impairment.
Time Frame: Baseline to Week 26
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | NB + CLI | Usual Care
Number analyzed (Participants) | 71 | 82
units on a scale | 16.4 (1.50) | -1.0 (1.41)
Statistical Analysis 1: Comparison: NB + CLI vs Usual Care; Test type: Superiority or Other; p < 0.0001, ANCOVA; Mean Difference (Net) = 17.4, 95% CI 2-sided [13.45 to 21.36]

ADVERSE EVENTS:
Time Frame: Day 1 through Week 78
Description: Only serious adverse events (SAE) and treatment-emergent adverse events (TEAE) leading to discontinuation from full participation were collected in this study.
  The 1% frequency threshold for reporting other adverse events is based on All Subjects (Entire Study) column.
Groups:
- NB + CLI (Controlled Treatment Period): Naltrexone SR 32 mg/Bupropion SR 360 mg/day (NB) with Comprehensive Lifestyle Intervention (CLI)
  NB: Naltrexone SR 32 mg/Bupropion SR 360 mg (NB) in combination tablets (daily dosage)
  CLI: The Comprehensive Lifestyle Intervention (CLI) program included telephone counseling, internet education, goal setting, and online tracking tools.
  The Controlled Treatment Period was from Day 1 to Week 26.
- Usual Care (Controlled Treatment Period): Usual Care (self-directed lifestyle intervention)
  Usual Care: Usual Care was a self-directed lifestyle intervention in which subjects were given calorie targets, instructions to increase exercise, and a pamphlet about weight loss by study site staff.
  The Controlled Treatment Period was from Day 1 to Week 26.
- All Subjects (Entire Study): Naltrexone SR 32 mg/Bupropion SR 360 mg/day (NB) with Comprehensive Lifestyle Intervention (CLI)
  NB: Naltrexone SR 32 mg/Bupropion SR 360 mg (NB) in combination tablets (daily dosage)
  CLI: The Comprehensive Lifestyle Intervention (CLI) program included telephone counseling, internet education, goal setting, and online tracking tools.
  All Subjects (Entire Study) consisted of all subjects in both the Controlled and Uncontrolled Treatment Periods. At the end of the Controlled Treatment Period (Week 26), subjects assigned to NB+CLI continued with NB+CLI for the duration of the study and subjects assigned to Usual Care were switched to NB+CLI for the duration of the study.
Arm/Group | NB + CLI (Controlled Treatment Period) | Usual Care (Controlled Treatment Period) | All Subjects (Entire Study)
Serious Adverse Events (participants affected / at risk) | 1/153 | 0/89 | 2/242
Other Adverse Events (participants affected / at risk) | 26/153 | 0/89 | 32/242
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | NB + CLI (Controlled Treatment Period) (N=153) | Usual Care (Controlled Treatment Period) (N=89) | All Subjects (Entire Study) (N=242)
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 2 (2) — One subject experienced an SAE during the Uncontrolled Treatment Period.
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | NB + CLI (Controlled Treatment Period) (N=153) | Usual Care (Controlled Treatment Period) (N=89) | All Subjects (Entire Study) (N=242)
Nausea (Gastrointestinal disorders) | 16 (16) | 0 (0) | 17 (17)
Anxiety (Psychiatric disorders) | 5 (5) | 0 (0) | 5 (5)
Headache (Nervous system disorders) | 2 (2) | 0 (0) | 4 (4)
Insomnia (Psychiatric disorders) | 2 (2) | 0 (0) | 3 (3)
Dizziness (Nervous system disorders) | 1 (1) | 0 (0) | 3 (3)
Constipation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 3 (3)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
If not already published by Sponsor as part of a multi-center publication, 24 months after conclusion, abandonment or termination of the study or notification that there will be no such multi-center publication, PI may publish the results for PI's study center individually. Prior to such publication, PI must provide Sponsor with at least 90 days to review and comment on the proposed publication. Sponsor may delay publication for up to an additional 6 month period to file for patent protection.